CLINICAL TRIAL: NCT04976452
Title: Identifying Learning Strategies to Improve Blood Pressure Measurement in Physical Therapy Education Programs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Youngstown State University (Other)
Collaborators: Midlothian Free Health Clinic (Unknown)
Responsible Party: Principal Investigator, Edmund Ickert, Assistant Professor, Youngstown State University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2021-122
Record Dates: First submitted 2021-07-15; First posted 2021-07-26 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Blood Pressure Measurement
Keywords: Physical Therapy; Teaching; Education

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Group 1 will include first year Physical Therapy students who will be trained for Blood Pressure (BP) measurement using a brief powerpoint lecture, completion of an interactive BP measurement module from the American Medical Association which includes a quiz assessment and certificate of completion, and a competency examination during the lab portion of class.
  Interventions: Other: Multi-component teaching content
- Group 2 (No Intervention): Group 2 consists of second year PT students who only had a powerpoint lecture on Blood Pressure measurement that was done virtually with no lab component or American Medical Association interactive module training.

INTERVENTIONS:
Other: Multi-component teaching content — The students assigned to Group 1 will undergo interactive module training by the American Medical Association which outlines how to properly measure blood pressure manually following the American Heart Association guidelines. Following completion of the module, students will be presented with a powerpoint lecture by the Primary Investigator on Blood Pressure. Students will then undergo a competency examination that assesses their ability to measure blood pressure following the guidelines of the American Heart Association.
  Other Names: American Medical Association Interactive Training Module with Quiz and Certificate; Powerpoint Lecture and Presentation on Blood Pressure; Competency Based Examination of Blood Pressure Measurement by Students
  Arms: Group 1

SUMMARY:
The purpose of this study is to determine an effective teaching strategy for Physical Therapy students in a Doctor of Physical Therapy (DPT) program that will produce consistent and accurate measuring of patient BP readings in the healthcare clinic according to the guidelines established by the AHA.

ELIGIBILITY:
This study is anticipated to have 40-45 students as participants that can vary in age range, but will mostly be centered around the 21-30 year old age range demographically. Doctor of Physical Therapy (DPT) students that are enrolled in the DPT program at Youngstown State will be recruited for this study, along with, patients who receive Physical Therapy services at the Midlothian Free Clinic. The participants will also come from both gender groups, with no exclusion criteria based on age and gender for this study.

Exclusion Criteria:

Group 1 Exclusion criteria (Experimental group):

1. Must be admitted to DPT program at Youngstown State University
2. Complete the Blood Pressure (BP) measure training module in the Clinical Skills Foundation
3. Pass the competency lab examination in Clinical Skills Foundation (> 80% score)

Group 2 Exclusion criteria (Control group):

1. Must be admitted to DPT program at Youngstown State University
2. Have not completed the BP training module (AMA) and competency lab examination in the Clinical Skills Foundation course

Patient Exclusion criteria:

1. Must be able to follow basic commands
2. Must be able to perform a transfer to multiple surfaces

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2021-12-16 (Actual)

PRIMARY OUTCOMES:
Competency Assessment Form | When the student is performing the blood pressure measurement which will span approximately 15-20 minutes
  This form was developed by the Primary Investigator to objectively measure a student's ability to take a manual blood pressure reading following the established guidelines of the American Heart Association.

SECONDARY OUTCOMES:
Pre-Measurement Student Survey | 10 minute survey given prior to participating in the study to both groups of students
  A survey will be provided for students to complete prior to measuring blood pressure in the clinic. The components of the survey will assess: basic information related to confidence in blood pressure measurements, prior training (before entering the Doctor of Physical Therapy program), and identification of overall strengths and weaknesses when conducting blood pressure measurements.
Post-Measurement Student Survey | 10 minute survey given following participation in the study to both groups of students
  A survey will be provided for students to complete after measuring blood pressure in the clinic. The components of the survey will assess: items for the student to self-reflect on their performance and identify how confident they were in the procedure they used to complete the blood pressure measurements, and overall self-identified strengths and weaknesses.

OTHER OUTCOMES:
Medical History Form | This will be completed by patients who will have their blood pressure measured by students. The estimated time frame for completion is 15 minutes
  A basic medical history form that identifies the patient's: past medical history, surgical history, and current medication use.
Post-Measurement Patient Survey | The is completed after blood pressure measurement and may take up to 15 minutes
  This is a survey that will be completed by patients after they have had their blood pressure measurement taken by the student. The items on this survey focus on: the patients confidence in the student's ability to perform their BP measurement, and qualitative feedback regarding both positive and negative aspects of student performance.

CONTACTS AND LOCATIONS:
Overall Officials: Edmund C Ickert, PT, DPT, MS, Principal Investigator — Youngstown State University
Locations (1):
- Midlothian Free Clinic, Youngstown, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Holmstrup M, Jensen B, Burkart R, Levis M. Using a novel assessment of procedural proficiency provides medical educators insight into blood pressure measurement. Int J Med Educ. 2016 Nov 19;7:375-381. doi: 10.5116/ijme.580b.2e4f. PMID 27864919
- [Background] Jaffe MG, Young JD. The Kaiser Permanente Northern California Story: Improving Hypertension Control From 44% to 90% in 13 Years (2000 to 2013). J Clin Hypertens (Greenwich). 2016 Apr;18(4):260-1. doi: 10.1111/jch.12803. Epub 2016 Mar 3. No abstract available. PMID 26939059
- [Background] Gordon CJ, Frotjold A, Fethney J, Green J, Hardy J, Maw M, Buckley T. The effectiveness of simulation-based blood pressure training in preregistration nursing students. Simul Healthc. 2013 Oct;8(5):335-40. doi: 10.1097/SIH.0b013e3182a15fa7. PMID 24061336
- [Background] Seybert AL, Barton CM. Simulation-based learning to teach blood pressure assessment to doctor of pharmacy students. Am J Pharm Educ. 2007 Jun 15;71(3):48. doi: 10.5688/aj710348. PMID 17619648
- [Background] Yamazaki Y, Hiyamizu I, Joyner K, Abe Y. Relation of clinical context to accuracy of simulator-based blood pressure measurement by first-year medical students. Int J Med Educ. 2018 Dec 21;9:325-331. doi: 10.5116/ijme.5c0f.935c. PMID 30589414
- [Background] Bland M, Ousey K. Preparing students to competently measure blood pressure in the real-world environment: a comparison between New Zealand and the United Kingdom. Nurse Educ Pract. 2012 Jan;12(1):28-35. doi: 10.1016/j.nepr.2011.04.009. Epub 2011 Jun 8. PMID 21641869
- [Background] Severin R, Wang E, Wielechowski A, Phillips SA. Outpatient Physical Therapist Attitudes Toward and Behaviors in Cardiovascular Disease Screening: A National Survey. Phys Ther. 2019 Jul 1;99(7):833-848. doi: 10.1093/ptj/pzz042. PMID 30883642
- [Background] Gazibara T, Rancic B, Maric G, Radovanovic S, Kisic-Tepavcevic D, Pekmezovic T. Medical students, do you know how to measure blood pressure correctly? Blood Press Monit. 2015 Feb;20(1):27-31. doi: 10.1097/MBP.0000000000000085. PMID 25243713
- [Background] Rakotz MK, Townsend RR, Yang J, Alpert BS, Heneghan KA, Wynia M, Wozniak GD. Medical students and measuring blood pressure: Results from the American Medical Association Blood Pressure Check Challenge. J Clin Hypertens (Greenwich). 2017 Jun;19(6):614-619. doi: 10.1111/jch.13018. Epub 2017 Apr 28. PMID 28452119
- [Background] Muntner P, Shimbo D, Carey RM, Charleston JB, Gaillard T, Misra S, Myers MG, Ogedegbe G, Schwartz JE, Townsend RR, Urbina EM, Viera AJ, White WB, Wright JT Jr. Measurement of Blood Pressure in Humans: A Scientific Statement From the American Heart Association. Hypertension. 2019 May;73(5):e35-e66. doi: 10.1161/HYP.0000000000000087. PMID 30827125
- [Background] Gonzalez-Lopez JJ, Gomez-Arnau Ramirez J, Torremocha Garcia R, Albelda Esteban S, Alio del Barrio J, Rodriguez-Artalejo F. Knowledge of correct blood pressure measurement procedures among medical and nursing students. Rev Esp Cardiol. 2009 May;62(5):568-71. doi: 10.1016/s1885-5857(09)71840-7. English, Spanish. PMID 19406072
- [Background] Crosley AM, Rose JR. Knowledge of accurate blood pressure measurement procedures in chiropractic students. J Chiropr Educ. 2013 Fall;27(2):152-7. doi: 10.7899/JCE-13-3. Epub 2013 Jun 27. PMID 23957320
- [Background] Ibiyemi O, Ogunbodede O, Gbolahan OO, Ogah OS. Knowledge and practices of blood pressure measurement among final year students, house officers, and resident dental surgeons in a dental hospital, South West Nigeria. Niger J Clin Pract. 2020 Jun;23(6):848-856. doi: 10.4103/njcp.njcp_416_19. PMID 32525122
- [Background] Arangalage D, Abtan J, Gaschignard J, Ceccaldi PF, Remini SA, Etienne I, Ruszniewski P, Plaisance P, De Lastours V, Lefort A, Faye A. Implementation of a large-scale simulation-based cardiovascular clinical examination course for undergraduate medical students - a pilot study. BMC Med Educ. 2019 Sep 18;19(1):361. doi: 10.1186/s12909-019-1750-4. PMID 31533700
- [Background] Chen JJ, Johannesmeyer HJ. Gagne's 9 Events of Instruction With Active Learning: Teaching Student Pharmacists How to Measure Blood Pressure. J Pharm Pract. 2021 Jun;34(3):407-416. doi: 10.1177/0897190019875610. Epub 2019 Sep 16. PMID 31526081
- [Background] Rabbia F, Testa E, Rabbia S, Pratico S, Colasanto C, Montersino F, Berra E, Covella M, Fulcheri C, Di Monaco S, Buffolo F, Totaro S, Veglio F. Effectiveness of blood pressure educational and evaluation program for the improvement of measurement accuracy among nurses. High Blood Press Cardiovasc Prev. 2013 Jun;20(2):77-80. doi: 10.1007/s40292-013-0012-5. Epub 2013 May 8. PMID 23653174
- [Background] Ballard G, Piper S, Stokes P. Effect of simulated learning on blood pressure measurement skills. Nurs Stand. 2012 Oct 24-30;27(8):43-7. doi: 10.7748/ns2012.10.27.8.43.c9363. PMID 23189601
- [Background] Leung GK, Nicholls JM. Effect of clinical context on simulator-based assessment of blood pressure taking - a pilot randomized study. Med Teach. 2014 Feb;36(2):177-9. doi: 10.3109/0142159X.2013.849328. Epub 2013 Oct 24. PMID 24156287
- [Background] Weber MA, Schiffrin EL, White WB, Mann S, Lindholm LH, Kenerson JG, Flack JM, Carter BL, Materson BJ, Ram CV, Cohen DL, Cadet JC, Jean-Charles RR, Taler S, Kountz D, Townsend RR, Chalmers J, Ramirez AJ, Bakris GL, Wang J, Schutte AE, Bisognano JD, Touyz RM, Sica D, Harrap SB. Clinical practice guidelines for the management of hypertension in the community: a statement by the American Society of Hypertension and the International Society of Hypertension. J Clin Hypertens (Greenwich). 2014 Jan;16(1):14-26. doi: 10.1111/jch.12237. Epub 2013 Dec 17. No abstract available. PMID 24341872
- [Background] Elliott KE, McCall KL, Fike DS, Polk J, Raehl C. Assessment of manual blood pressure and heart rate measurement skills of pharmacy students: a follow-up investigation. Am J Pharm Educ. 2008 Jun 15;72(3):60. doi: 10.5688/aj720360. PMID 18698382
- [Background] Yamazaki Y, Hiyamizu I, Joyner K, Otaki J, Abe Y. Assessment of blood pressure measurement skills in second-year medical students after ongoing simulation-based education and practice. Med Educ Online. 2021 Dec;26(1):1841982. doi: 10.1080/10872981.2020.1841982. PMID 33135567
- [Background] Leong C, Louizos C, Frankel G, Ng S, Iacovides H, Falk J, Dunford D, Brink K, Kleiman N, Davis C, Renaud R. A physical assessment skills module on vital signs. Am J Pharm Educ. 2014 Sep 15;78(7):137. doi: 10.5688/ajpe787137. PMID 25258442
- [Background] Grim CM, Grim CE. A curriculum for the training and certification of blood pressure measurement for health care providers. Can J Cardiol. 1995 Nov;11 Suppl H:38H-42H. PMID 7489543